CLINICAL TRIAL: NCT04860934
Title: Efficacy Of Dual Task Training On Children With Ataxia After Medulloblastoma Resection
Brief Title: Dual Task Training On Children With Ataxia After Medulloblastoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHE-BT004
Record Dates: First submitted 2021-03-21; First posted 2021-04-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Medulloblastoma, Childhood; Childhood Cancer
Keywords: Ataxia; Medulloblastoma Resection; posterior fossa tumor; physical activity; Dual Task Training; Childhood Cancer
MeSH Terms: conditions — Medulloblastoma; Neoplasms; Ataxia; Infratentorial Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental controlled randomization using Block Stratified Randomized Software program, after obtaining informed consent from illegible patient or his caregiver.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy (Active Comparator): Each child in this group will receive the selected physical therapy program which include mobility exercises, strengthening exercises, balance exercises, gait training exercises, and exercises to improve physical conditioning for one-hour session three times weekly for 8 successive weeks
  Interventions: Behavioral: Control Group
- Physical therapy + Dual Task Training Program (Experimental): Each child in this group will perform one-hour session consist of two tasks (cognitive and balance task) in addition to the selected physical therapy program as control group three times weekly for 8 successive weeks.
  Interventions: Behavioral: Dual Task Training Program Group; Behavioral: Control Group

INTERVENTIONS:
Behavioral: Dual Task Training Program Group — Fifteen patients will receive Dual Task Training Program. Total Period: 8 Weeks.
  Arms: Physical therapy + Dual Task Training Program
Behavioral: Control Group — Each child in this group will receive the selected physical therapy program which include mobility exercises, strengthening exercises, balance exercises, gait training exercises, and exercises to improve physical conditioning for one-hour session three times weekly for 8 successive weeks.

SUMMARY:
Medulloblastoma is a rapidly-growing tumor of the cerebellum, this area controls balance, posture and sophisticated motor functions like finer hand movements, speech, and swallowing. With the goal of, complete resection, major complications during tumor removal are usually caused by damage to the brain stem and injury to the lower cranial nerves.It has been reported that those children present Ataxia after resection. So the purpose of this study is to investigate the effectiveness of using a selected dual-task- training program to improve postural stability in those Children.

DETAILED DESCRIPTION:
Most patients present with symptoms of hydrocephalus due to obstruction by tumor at the level of the fourth ventricle or cerebral aqueduct, and ataxia (Martin et al., 2014). If the tumor is large enough, the lesion itself can also cause mass effect and increased intracranial pressure. Furthermore, direct structural damage from the children can thus present with nausea, vomiting, ataxia,diplopia.

Ataxia in children is a common clinical sign of various origins consisting of impaired coordination of movement and balance with a lack of muscle control during voluntary activity. Ataxia is most frequently caused by dysfunction of the complex circuitry connecting the basal ganglia, cerebellum and cerebral cortex, and this type of involvement is recorded as "cerebellar ataxia.

Recently, the evidence for procedural memory training has advanced sophistication to suggest and ultimately prove that automaticity of a primary (motor task can be developed through exposure to massive repetitions practice) and the forced subconscious processing using dual task interference (Bermúdez, 2017).

The Objectives of the Study:

1- Aim of the Study: Determining the efficacy of "Dual Task Training in children with ataxia after Medulloblastoma Resection regarding "Static Balance" and "Dynamic Balance" as indicators of Postural Control

2-Specific Objectives:

1. Assess static balance by measuring center of pressure using force plate mode in the humac balance system.
2. Assess dynamic balance by using tilt mode in the humac balance system .
3. Evaluate the improvement on functional status and independence in ADL activities by functional independence measurement.
4. Determine the more effective program for rehabilitation of children with ataxia

3-Secondary Objectives:

1. Assess the degree of ataxia in children after medulloblastoma resection by SARA scale.
2. Detect the effect of cognitive interference on postural stability and balance.
3. Detect if there is improvement in cognitve function after dual task training.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from (5-10 years).
2. Severity of ataxia will be from 15-30 by SARA scale.
3. Children after 2 months of medulloblastoma resection.
4. They can stand and walk with minimal support.
5. They have good cognition, compliance, and ability to understand and execute test instructions.
6. Children receiving radiotherapy and chemotherapy sessions
7. They are medically stable

Exclusion Criteria:

Children will be excluded from the study if they have

1. Any neuromuscular disorder.
2. Visual impairment.
3. Cognitive problem
4. Convulsion.
5. Peripheral neuropathy due to chemotherapy.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Dual Task Training program | 8 Weeks
  Determining the efficacy of "Dual-Task Training in children with ataxia after Medulloblastoma Resection regarding "Static Balance" and "Dynamic Balance" will be assessed with HUMAC Balance system as indicators of Postural Control

SECONDARY OUTCOMES:
Ataxia after Medulloblastoma Resection | 8 Weeks
  The degree of ataxia will be assessed in children by SARA (Scale of Assessment and Rating of Ataxia) with a scoring scale with minimum value (0, which means there is no Ataxia) and maximum values (40, high score of Ataxia).

OTHER OUTCOMES:
Balance system in children with ataxia after Medulloblastoma Resection | 8 Weeks
  Will be assessed with Pediactris Balance Scale with scoring range with a scoring scale with minimum value (0, which means the child has no balance ) and maximum values (56, which means the child has a good balance score).
ADL (activity of daily living) in children with ataxia after Medulloblastoma Resection | 8 Weeks
  assessment of ADL (activity of daily living) with functional independence measurement questionnaire which the higher scores mean a better daily activity independence lower score means worse activity with dependency in function.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mostafa Sedeek, BSc, Principal Investigator — Cairo University
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt

REFERENCES:
- [Derived] Selim FM, Elshafey MA, El-Ayadi MM, Albeltagi DM, Ali MS. Efficacy of dual-task training on stability and function in children with ataxia after medulloblastoma resection: A randomized controlled trial. Pediatr Blood Cancer. 2023 Nov;70(11):e30613. doi: 10.1002/pbc.30613. Epub 2023 Aug 10. PMID 37561355